CLINICAL TRIAL: NCT02889341
Title: Valuation of Variable Dose of Docosahexanoic Acid for the Improvement of the Parameters of Male Fertility
Acronym: DHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1303-SEV-00-CG
Record Dates: First submitted 2016-08-04; First posted 2016-09-05 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2016-12

CONDITIONS: Male Infertility
Keywords: Docosahexanoic Acid,; DNA fragmentation; male fertility; Sperm parameters improvements
MeSH Terms: conditions — Infertility, Male | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 500 mg DHA/day (Active Comparator): 500 mg DHA/day
  Interventions: Dietary Supplement: DHA
- 1g DHA/day (Active Comparator): 1g DHA/day
  Interventions: Dietary Supplement: DHA
- 2g DHA/day (Active Comparator): 2g DHA/day
  Interventions: Dietary Supplement: DHA

INTERVENTIONS:
Dietary Supplement: DHA
  Other Names: Docosahexaenoic acid
  Arms: 1g DHA/day; 2g DHA/day; 500 mg DHA/day
Other: Placebo
  Arms: Placebo

SUMMARY:
Sperm parameters will be examined before DHA (DHA=Docosahexanoic Acid) consumption, after one months and after 2 months taken Docosahexanoic Acid or placebo.

DETAILED DESCRIPTION:
Prospective, randomized, double blind, placebo-controlled intervention study within individuals. Assisted reproduction unit and academic research laboratory. One hundred an eighty human semen samples from 60 infertile patients of IVI Sevilla clinic were finally included. Assessment of oxidative stress, apoptosis, lipid peroxidation, mitochondrial membrane potential, DNA fragmentation and standard sperm parameters before and after supplementation with different DHA doses (0.5, 1 and 2 g) or placebo for 1 and 3 months.

ELIGIBILITY:
Inclusion criteria:

* 1 year of infertility
* > 10 mill/ml of sperms
* Motility < 60% progressive
* Morphology < 2% (WHO 2010)

Exclusion criteria:

No meeting the inclusion criteria.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sperm cell concentration | Three months
  Measured in millions of sperm cells per ml of semen sample
Sperm cell motility | Three months
  Measured in percentage of each type of motile sperm according to OMS 2010 criteria (A-D).
Sperm cell morphology | Three
  Measured in percentage of sperm cell with normal morphology according to OMS 2010 criteria.

IPD SHARING:
Plan to Share IPD: No